CLINICAL TRIAL: NCT07175259
Title: Relation of Total Ischemic Time to Repolarization Indices and Their Impact on Outcomes Among STEMI Patients Undergoing Primary PCI
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Monazea Menisy Khaled, Principal Investigator, Assiut University
Other Study IDs: Repolarization indices PPCI
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: ST Elevation (STEMI) Myocardial Infarction of Other Sites; Repolarization Indices; Total Ischemic Time; Primary Percutaneous Coronary Intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Echocardiography — Simple, bedsides, non invasive

SUMMARY:
1. Evaluate The impact of early versus late presentation on electrocardiographic ventricular repolarization indices.
2. To assess the association between repolarization indices among early, late presentation in relation to in-hospital ventricular arrhythmias, in-hospital MACE, and 6 months MACE.

DETAILED DESCRIPTION:
ST-elevation myocardial infarction (STEMI) remains a time-critical cardiovascular emergency. Early reperfusion is essential to reduce myocardial necrosis, preserve ventricular function, and improve survival outcomes. However, delayed presentation remains a significant problem, especially in developing countries, leading to larger infarct sizes and worse clinical outcomes. (Park J, Choi KH, Lee JM, et al. 2019) Ventricular repolarization indices including QT interval ( Measured from the onset of the QRS complex (beginning of Q wave or R if no Q visible)To the end of the T wave returning to the isoelectric line ), QT dispersion (QTD) ( Calculated as: QTD = QT{max} - QT{min}), corrected QT interval (QTc) Calculated using Bazett's formula: QTc = {QT}/{sqrt{RR}. Corrected QT dispersion (cQTD or QTcd) Calculated as: cQTD = QTc{max}- QTc{min}.TPE/QT ratio, Calculated as: {TPE/QT Ratio} = {TPE}/{QT}, T peak-to-Tend interval (TPE) ( Measured from the peak of the T wave To the end of the T wave returning to the isoelectric line ), are non-invasive markers of electrical instability and myocardial injury. Prolongation of these indices has been associated with worse microvascular perfusion (including the no-reflow phenomenon (Abdelmeguid AE, Abdelhamid SM, Abdelhameed KM, et al. 2023) and lower myocardial blush grade [MBG]) (Liu X, Li Y, Li D, et al. 2021) and higher rates of major adverse cardiovascular events (MACE). (Çağdaş M, Rencüzoğulları İ, Karakoyun S, et al. 2018, Abdelmeguid AE, Abdelhamid SM, Abdelhameed KM, et al. 2023, Liu X, Li Y, Li D, et al. 2021) There is limited data assessing the direct relationship between early vs late presentation, repolarization indices measured before and after PCI, and subsequent outcomes in STEMI patients, particularly in our local population.

This study aims to fill this gap by investigating whether timing of presentation significantly affects repolarization indices and whether these indices can predict in-hospital and six-month clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

- Patients presenting with acute STEMI undergoing primary PCI

Exclusion Criteria:

- 1. Prior myocardial infarction or CABG. 2. Left or right bundle branch block. 3. Atrial fibrillation. 4. Cardiac arrest or cardiogenic shock 5. Valvular heart disease (severe). 6. Use of QT-prolonging medications as anti-arrhythmic, anti-psychotic, anti-depressant and some types of antibiotics.

7. Poor quality ECG tracings. 8. Chronic kidney disease stage ≥3. 9. Electrolyte abnormalities at admission 10. Undetermined date of pain

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include patients presenting with ST-elevation myocardial infarction (STEMI) who are admitted to the coronary care unit and undergo primary percutaneous coronary intervention (PCI) as the reperfusion strategy. Eligible patients will be adults presenting within the accepted therapeutic window for primary PCI.
  The final sample will thus represent a consecutive cohort of STEMI patients undergoing primary PCI, allowing assessment of the relationship between total ischemic time and repolarization indices (QTc, Tpe interval, Tpe/QT ratio, etc.), and their subsequent impact on both short- and long-term clinical outcomes.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Association between total ischemic time and ventricular repolarization indices | 6 months
  Correlation between total ischemic time (symptom onset to balloon time) and ECG-derived repolarization parameters, including QT interval, corrected QT (QTc), Tpeak-Tend interval, and Tpeak-Tend/QT ratio. Analysis will evaluate linear correlations and threshold effects.

SECONDARY OUTCOMES:
In-hospital ventricular arrhythmias | 7 dayes
  Occurrence of sustained ventricular tachycardia or ventricular fibrillation documented during index hospitalization.
In-hospital major adverse cardiovascular events (MACE) | 7 days
  Composite of all-cause death, reinfarction (per universal definition of MI), and new or worsening heart failure during index hospitalization.
Six-month major adverse cardiovascular events (MACE) | 6 months
  Composite of cardiovascular mortality, hospitalization for heart failure or recurrent ACS, and target lesion revascularization (TLR) at follow-up.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang X, Zhang L, Gao C, Zhu J, Yang X. Tpeak-Tend/QT interval predicts ST-segment resolution and major adverse cardiac events in acute ST-segment elevation myocardial infarction patients undergoing percutaneous coronary intervention. Medicine (Baltimore). 2018 Oct;97(43):e12943. doi: 10.1097/MD.0000000000012943. PMID 30412109
- [Background] Rao SV, O'Donoghue ML, Ruel M, Rab T, Tamis-Holland JE, Alexander JH, Baber U, Baker H, Cohen MG, Cruz-Ruiz M, Davis LL, de Lemos JA, DeWald TA, Elgendy IY, Feldman DN, Goyal A, Isiadinso I, Menon V, Morrow DA, Mukherjee D, Platz E, Promes SB, Sandner S, Sandoval Y, Schunder R, Shah B, Stopyra JP, Talbot AW, Taub PR, Williams MS. 2025 ACC/AHA/ACEP/NAEMSP/SCAI Guideline for the Management of Patients With Acute Coronary Syndromes: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2025 Apr;151(13):e771-e862. doi: 10.1161/CIR.0000000000001309. Epub 2025 Feb 27. PMID 40014670
- [Background] Demidova MM, Carlson J, Erlinge D, Azarov JE, Platonov PG. Prolonged Tpeak-Tend interval is associated with ventricular fibrillation during reperfusion in ST-elevation myocardial infarction. Int J Cardiol. 2019 Apr 1;280:80-83. doi: 10.1016/j.ijcard.2019.01.008. Epub 2019 Jan 4. PMID 30661844
- [Background] Abu Shajahan M, Mohideen B, P A J, Thaha SM, Ashraf AR, Nazar I, Nair RG, Fakhrudeen Mushthak S, Suresh AL. Prognostic Value of QTc Dispersion in Acute Myocardial Infarction. Cureus. 2025 Apr 23;17(4):e82846. doi: 10.7759/cureus.82846. eCollection 2025 Apr. PMID 40416232
- [Background] Cagdas M, Karakoyun S, Rencuzogullari I, Karabag Y, Yesin M, Uluganyan M, Gursoy MO, Artac I, Ilis D, Efe SC, Tasar O. Relationship between R-wave peak time and no-reflow in ST elevation myocardial infarction treated with a primary percutaneous coronary intervention. Coron Artery Dis. 2017 Jun;28(4):326-331. doi: 10.1097/MCA.0000000000000477. PMID 28207567